CLINICAL TRIAL: NCT00306514
Title: A Phase IIa Study to Evaluate Safety, Tolerability, and Immunogenicity of a Melan-A VLP Vaccine in HLA-A2 Positive Patients With Stage III/IV Malignant Melanoma
Brief Title: Safety and Immunogenicity of a Melan-A VLP Vaccine in Advanced Stage Melanoma Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cytos Biotechnology AG (Industry)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: CYT004-MelQbG10 01
Record Dates: First submitted 2006-03-23; First posted 2006-03-24 (Estimated); Last update posted 2007-09-20 (Estimated); Status verified 2007-09

CONDITIONS: Melanoma
Keywords: metastatic malignant melanoma of the skin
MeSH Terms: conditions — Melanoma

INTERVENTIONS:
Biological: CYT004-MelQbG10

SUMMARY:
The purpose of this study is to evaluate whether vaccination with a Melan-A VLP vaccine leads to a specific cellular immune response in patients with malignant melanoma at advanced stage of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent
* Able and willing to complete all protocol requirements
* Age: 18 years and older
* Histologically confirmed stage III or IV melanoma
* HLA-A*0201 haplotype
* Expected survival of at least 6 months
* ECOG performance status of 0 or 1
* At least one and no more than 2 previous systemic therapies for metastatic melanoma
* Able to undergo computed tomography (CT) scan/ magnetic resonance imaging (MRI) scan for tumor assessment.
* Lack of response to or progression after most recent systemic therapy for metastatic melanoma.
* Adequate organ and bone marrow functions
* All adverse events (AEs) from prior anticancer therapy have resolved to ≤ Grade 1
* Sexually active males should use adequate contraception throughout the study period and 3 months thereafter.
* Females of child bearing potential should use adequate contraception throughout the study period and 3 months thereafter, that can be oral contraception or a double-barrier local contraception (intra-uterine device plus condom or spermicidal gel plus condom), and have a negative serum pregnancy test within 4 weeks prior to the first dose of the vaccine.

Exclusion Criteria:

* Pregnant or nursing
* Use of an investigational drug within 30 days before enrollment
* Known or suspected brain metastases
* Active malignancy in the 5 years prior to enrollment other than melanoma, basal cell carcinoma or cervical carcinoma in situ.
* Major surgery within 4 weeks prior to enrollment.
* Current use of an immunosuppressive drug or any concomitant medication that could potentially interfere with the study drug.
* Presence of significant cardiovascular, renal, pulmonary, endocrine, infectious, or neurological disorders.
* Serum tests positive for HIV, hepatitis B virus (HBV), hepatitis C virus (HCV).
* Active autoimmune diseases or severe allergies.
* Known type 1 allergy.
* Current diagnosis or history of relevant and severe psychiatric disorder that compromises the patient's ability to understand the patient information, to give informed consent, to comply with the trial protocol or to complete the study.
* Blood donation or loss of > 400mL within 8 weeks prior to inclusion.
* Hemoglobin (Hb) < 10g/dL
* Abuse of alcohol or other recreational drugs.
* Previous vaccination with a Melan-A peptide analogue.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Wolfram Sterry, MD, Principal Investigator — University Hospital Charite, Berlin, D
Locations (1):
- Dept. of Dermatology, Venerology and Allergy, Berlin, State of Berlin, Germany